CLINICAL TRIAL: NCT03509090
Title: Evaluation of the Analgesic Efficacy of Ultrasound-guided Erector Spinae Block in Unilateral Breast Cancer Surgery: Randomized Controled Study.
Brief Title: Erector Spinae Block in Segmental Mastectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Onur Selvi, MD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-AKD-186
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: regional anesthesia; erector spinae plane block; postoperative pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): Unilateral ESP block will be applied as postoperative regional analgesia technique in addition to the multimodal therapy. Then she is positioned in a right lateral position to perform ESP blocks. The skin will be disinfected and ESP block at one side will be performed in the lateral decubitus position and at T4 transverse process level by using 10-MHz linear ultrasound probe (Logic Ebook XP General Electrics, USA). The probe will be located 3 cm lateral to T4 spinous process in longitudinal parasagittal orientation. An 8 cm 21 gauge needle (BRAUN Stimuplex A®, Germany) will be inserted by using out of the plane technique. The ESP blocks proceed with 15 ml of 0,25% bupivacaine, 7,5 ml 1 % lidocaine, ,7,5 ml 0,9 % NaCl as total 30 ml . The injections will be applied after the confirmation of location by hidrodisection developed anterior to erector spinae muscle with 1-2 ml of local anesthetic solution.
  Interventions: Procedure: erector spinae block
- Control group (Active Comparator): In this group, patients will receive only multimodal analgesic treatment including patient-controlled analgesia prepared with tramadol. Patient-controlled analgesia (PCA) with tramadol at 3mg/cc concentration is programmed with no basal infusion, demand dose 10 mg and 20-minute lock-out interval. Also, patients received 1 gr paracetamol in every 6 hours.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: erector spinae block — erector spinae block will be performed in this group as postoperative analgesia treatment.
  Arms: ESP block group
Procedure: Control group — patients will receive only multimodal analgesic treatment including patient-controlled analgesia
  Arms: Control group

SUMMARY:
Erector spinae plane block (ESPB) is a recently described block. Although there is still no consensus of its mechanism, the published case series seems to promise a new regional anesthesia technique for both chronic and acute pain. In this clinical trial, the postoperative analgesic effect of ESPB will be studied in patients underwent unilateral breast cancer surgery.

DETAILED DESCRIPTION:
In this study 30 patients will be enrolled to study between March 2018-August 2018. All patient will be randomly selected who will be operated for breast cancer surgery between determined dates. Age, weight, ASA score, body mass index , additional dissease ststus will be recorded. The patients will be divided in two groups. One group will have ESPB at the end of the operation and the second group will be treated with multimodal analgesia techniques and both groups will receive patient controlled analgesia. Both groups will receive identical anaethesia protocols. Perioperative analgesia protocols will provide acetaminophen 1 gr and the same dose will be repeated in every 6 hours regardless of the pain scores. In postoperative period the pain scores of the patients will be recorded according to the numeric rating scale (NRS) in every three hours. If pain score raises over 4/10 on NRS the patient will receive tramadol 100mg as rescue analgesia. In case of persisting pain first, meperidine 50 mg will be apllied and other multimodal analgesic drugs will be added to protocol. At the end of the study 24 hours total opioid usage of patients, pain scores and side effects will statistically be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Being volunteer
2. Over 18 years old
3. Unilateral segmental mastectomy patients

Exclusion Criteria:

1. Emergency operations
2. Younger than 18 years old,
3. Non Volunteers
4. ASA 3 and 4 patients
5. Non-cooperative patients

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
postoperative anaglesic effect of ESPB in unilateral segmental mastectomy patients | 24 hours postoperatively
  Post operative pain scores will be recorded with NRS and opioid usage will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Result] Bonvicini D, Giacomazzi A, Pizzirani E. Use of the ultrasound-guided erector spinae plane block in breast surgery. Minerva Anestesiol. 2017 Oct;83(10):1111-1112. doi: 10.23736/S0375-9393.17.12015-8. Epub 2017 May 11. No abstract available. PMID 28492298